CLINICAL TRIAL: NCT06350487
Title: The Efficacy of Enavogliflozin on Exercise Performance and Diastolic Function in Heart Failure With Preserved Ejection Fraction: A Randomized Controlled Trial
Brief Title: The Efficacy of Enavogliflozin in Heart Failure With Preserved Ejection Fraction
Acronym: ENRICH-PEF
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeong Hoon Yang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SMC2024-01-089-003
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure, Preserved Ejection Fraction
Keywords: Heart failure with preserved ejection fraction; Sodium glucose cotransporter 2 inhibitors; Exercise performance
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Intervention Model Description: A prospective, open label, single center, randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: Clinical outcome assessment will be performed under blinded assessment about the allocated treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGLT2 inhibitor group (Experimental): SGLT2 inhibitor group will receive Enavogliflozin (0.3mg oral tablet once daily).
  Interventions: Drug: SGLT2 inhibitor
- Control group (No Intervention): Control group will not receive any SGLT2 inhibitors during the study period.

INTERVENTIONS:
Drug: SGLT2 inhibitor — Enavogliflozin (0.3mg oral tablet once daily) will be administrated.
  Other Names: SGLT2 inhibitor: Enavogliflozin (Brand names: Envlo tab)
  Arms: SGLT2 inhibitor group

SUMMARY:
The aim of prospective, open label, single center, randomized controlled trial is to investigate the efficacy of enavogliflozin on exercise performance, diastolic dysfunction, and quality of life in patients with heart failure with preserved ejection fraction (HFpEF).

DETAILED DESCRIPTION:
HFpEF is a clinically heterogenous syndrome and has unique characteristics that differ from the other entities of heart failure. Cardiovascular and non-cardiovascular comorbidities are known to contribute to the pathogenesis of HFpEF, and consequently, the importance of HFpEF is increasingly emphasized as the population ages. In fact, HFpEF occurs in approximately 5% of the general population aged over 60 years and account for half of hospitalization for heart failure. Notwithstanding, no medication has been found to be effective for HFpEF. Only recently, Sodium glucose cotransporter 2 (SGLT2) inhibitors was proven effective in patients with HFpEF in two landmark trials, EMPEROR-Preserved and DELIVER trials. In both trials, SGLT2 inhibitor was consistently associated with reduced risk of composite outcome of cardiovascular death and hospitalization for heart failure. In this regard, 2023 focused update of the 2021 European Society of Cardiology (ESC) guidelines for heart failure recommends SGLT2 inhibitor as class 1A recommendation in patients with HFpEF.

Despite the solid evidence about the clinical benefit of SGLT2 inhibitor in patients with HFpEF, little is known about the mechanisms responsible for the beneficial cardiac effects of SGLT2 inhibitor. Patients with HFpEF are known to have impaired exercise and functional capacity, which lead to declined quality of life and debilitating symptoms. Along with unclear mechanisms responsible for the beneficial cardiac effect of SGLT2 inhibitor, the impacts of SGLT2 inhibitor on exercise and functional capacity in patients with HFpEF have also not been clearly evaluated. Therefore, this trial aim to evaluate the impact of SGLT2 inhibitor on exercise performance, diastolic function, and quality of life in patients with HFpEF using newly developed SGLT2 inhibitor, Enavogliflozin.

ELIGIBILITY:
1. Inclusion Criteria:

1) Age ≥19 2) New York Heart Association (NYHA) II-III dyspnea 3) Diagnosis of HFpEF (Exams conducted within 6 months from screening) [must satisfy all (1), (2), and (3)]

1. Left ventricular ejection fraction (LVEF) ≥50%
2. NT-proBNP ≥220 pg/mL or BNP ≥80 pg/mL, if in sinus rhythm NT-proBNP ≥660 pg/mL or BNP ≥240 pg/mL, if in atrial fibrillation
3. Satisfying either noninvasive or invasive criteria I. Noninvasive: Echocardiography with at least one of the following criteria

   * LAVI ≥34 ml/m2
   * Lateral E/e' ≥9
   * LVMI ≥115 g/m2 if male or ≥95 g/m2 if female
   * LV wall thickness ≥12mm II. Invasive: LVEDP ≥16mmHg or pulmonary capillary wedge pressure(PCWP) ≥15mmHg 4) Stable/chronic ambulatory patients without hospitalization within the last 30 days due to heart failure decompensation episode 5) Patients taking heart failure medication without change for at least 3 weeks before screening

     2. Exclusion Criteria:
     1. Unwillingness or inability to comply with the procedures described in this protocol
     2. The ability to walk is, in the investigator's opinion, clearly limited by joint disease or other locomotor problems or lung diseases rather than by cardiorespiratory fitness
     3. NYHA IV dyspnea
     4. Type 1 diabetes mellitus
     5. Estimated glomerular filtration rate (eGFR) <60 ml/min/1.73m2 (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula)
     6. Anemia (Hb <7g/dL)
     7. Severe hepatic impairment (Child-Pugh class C)
     8. Acute myocardial infarction or unstable angina within 30 days before inclusion or planned coronary revascularization at the time of inclusion
     9. Significant left-sided valvular heart disease (moderate to severe stenosis and severe regurgitation)
     10. Heart failure due to any of the following: infiltrative cardiomyopathy (amyloidosis, sarcoidosis), active myocarditis, constrictive pericarditis, hypertrophic cardiomyopathy
     11. Symptomatic hypotension (systolic blood pressure <90mmHg)
     12. Severe chronic obstructive pulmonary disease (postbronchodilator forced expiratory volume in 1 second (FEV1)/forced vital capacity(FVC) <70% and FEV1 <50%)
     13. Treated with sodium-glucose cotransporter-2 inhibitors (SGLT2i) within 30 days before inclusion
     14. History of diabetic ketoacidosis while in treatment with SGLT2i
     15. Recurrent genitourinary tract infections
     16. History of Hypersensitivity reaction to SGLT2i
     17. Non-cardiac co-morbid conditions are present with life expectancy <2 year or that may result in protocol non-compliance (per site investigator's medical judgment)
     18. Female patients who are currently or planning to become pregnant
     19. Female patients who are lactating
     20. Patients participating in other clinical trials

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in peak oxygen consumption (VO2) | Week 24
  Change in peak oxygen consumption (VO2) from baseline to week 24

SECONDARY OUTCOMES:
Change in minute ventilation to carbon dioxide output ratio (VE/VCO2 slope) | Week 24
  Change in minute ventilation to carbon dioxide output ratio (VE/VCO2 slope) from baseline to week 24
Change in Left atrial volume index (LAVI) before and after maximal exercise | Week 24
  Change in LAVI before and after maximal exercise from baseline to week 24
Change in Lateral Early diastolic transmitral filling velocity over early diastolic relaxation velocity at mitral annulus (E/e') before and after maximal exercise | Week 24
  Change in Lateral E/e' before and after maximal exercise from baseline to week 24
Change in Left ventricular mass index (LVMI) before and after maximal exercise | Week 24
  Change in LVMI before and after maximal exercise from baseline to week 24
Change in LV wall thickness before and after maximal exercise | Week 24
  Change in LV wall thickness before and after maximal exercise from baseline to week 24
Change in LV global longitudinal strain before and after maximal exercise | Week 24
  Change in LV global longitudinal strain before and after maximal exercise from baseline to week 24
Change in LA strain before and after maximal exercise | Week 24
  Change in LA strain before and after maximal exercise from baseline to week 24
Change in right ventricular (RV) free wall strain before and after maximal exercise | Week 24
  Change in RV free wall strain before and after maximal exercise from baseline to week 24
Change in health-related quality of life assessed by the Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CS) | Week 24
  Change in health-related quality of life assessed by the Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CS) from baseline to week 24
  Score ranges from 0 to 100 and higher value represents better quality of life.
Change in N-Terminal pro-B-type Natriuretic Peptide (NT-proBNP) level | Week 24
  Change in NT-proBNP level from baseline to week 24
Change in chronotropic response reserve assessed by change in heart rate from rest to peak exercise | Week 24
  Change in chronotropic response reserve assessed by change in heart rate from rest to peak exercise from baseline to week 24
Change in serum iron | Week 24
  Change in serum iron from baseline to week 24
Change in ferritin | Week 24
  Change in ferritin from baseline to week 24
Change in total iron binding capacity | Week 24
  Change in total iron binding capacity from baseline to week 24
Change in hemoglobin | Week 24
  Change in hemoglobin from baseline to week 24
All-cause death | Week 24
  All-cause death
Hospitalization for heart failure | Week 24
  Hospitalization for heart failure should include all of the following criteria:
  1. Hospitalization with primary diagnosis of heart failure
  2. Duration of hospitalization of at least 12 hours
  3. New or worsening symptoms of heart failure
  4. Objective evidence of new or worsening heart failure on physical examination or laboratory findings
  5. Initiation or intensification of heart failure treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hoon Yang, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, de-identified data will be shared upon reasonable request and with permission from the principal investigator.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication of first manuscript and trial results, de-identified data will be shared upon reasonable request and with permission from the principal investigator.
Access Criteria: After publication of first manuscript and trial results, de-identified data will be shared upon reasonable request and with permission from the principal investigator.